CLINICAL TRIAL: NCT01705587
Title: Fracture (FX) Improvement With Teriparatide: FiX-IT Study
Acronym: FiX-IT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Susan L. Greenspan (Other)
Collaborators: University of Pittsburgh (Other); Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Susan L. Greenspan, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO12040560 (FiX-IT)
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Osteoporosis; Atypical Femoral Fracture
Keywords: osteoporosis; atypical femoral fractures; prior bisphosphonate treatment; postmenopausal women; bone loss
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate teriparatide (Experimental): Open label teriparatide given immediately following surgical repair of fracture
  Interventions: Drug: teriparatide
- Delayed teriparatide (Experimental): Open label teriparatide given six months following surgical repair of fracture
  Interventions: Drug: teriparatide

INTERVENTIONS:
Drug: teriparatide — 20 microgram once-daily subcutaneous injection
  Other Names: Forteo

SUMMARY:
This open label comparison study examines the hypothesis that teriparatide given immediately following repair of an atypical subtrochanteric or diaphyseal femoral shaft fracture will enhance healing and improve bone mineral density compared to delayed treatment (after six months) with teriparatide or no treatment with teriparatide (patients who refuse therapy or for whom teriparatide is contraindicated). Patients with up-front teriparatide in addition will have greater quality of life measures and less pain compared to those with delayed or no therapy.

DETAILED DESCRIPTION:
Up to 24 postmenopausal women with osteoporosis who have been on bisphosphonate therapy for one year or more at any point prior to fracture and have sustained an atypical subtrochanteric or diaphyseal fracture will be enrolled. Subjects randomized to the two intervention arms will self-administer a daily SQ injection of the study medication for 12 months. The primary objective is to demonstrate greater radiologic evidence of healing at 10 weeks in patients on immediate teriparatide compared to those on delayed teriparatide who receive therapy six months after fracture. Secondary end points include (1) radiologic healing at 2, 6, 24, and 46 weeks; (2) increased bone density at 6 and 12 months as assessed by dual x-ray absorptiometry (DXA) at the spine, contralateral hip, and femoral neck; (3) quality of life improvements at 10 weeks and 6 months as assessed by quality of life questionnaire and pain score; and (4) differences in biochemical markers of bone turnover in patient with upfront therapy compared to patients with delayed therapy and patients who refuse therapy or for whom teriparatide is contraindicated.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women
* with osteoporosis who have been on bisphosphonate therapy for one year or more (all bisphosphonates will be included such as alendronate, risdedronate, ibandronate, or zoledronic acid).
* Patients will also be included if they are on glucocorticoids or other medications known to affect bone mineral metabolism as these are often found in patients with these types of fractures.
* sustain an atypical subtrochanteric or diaphyseal femoral shaft fracture as defined by the the 2010 ASBMR task force. An atypical fracture must include all of the following: (1) a location in the femur distal to lesser trochanter; (2) no trauma or minimal trauma as a fall; (3) transverse or short oblique configuration; (4) noncomminuted; and (5) complete fracture extends through both cortices and may be associated with a medial spike; incomplete fractures involve only the lateral cortex. Patients who have an incomplete fracture can be included if they fall into the 2010 ASBMR task force definition.

Exclusion Criteria:

* men
* children
* those who have had radiation therapy
* Paget's disease
* treatment with teriparatide for two year in the past
* metastatic bone disease
* active cancer
* hypercalcemia
* hyperparathyroidism
* metabolic disease other than osteoporosis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L. Greenspan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Osteoporosis Prevention & Treatment Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Teriparatide | Delayed Teriparatide
Started | 7 | 6
Completed | 7 | 5
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Teriparatide | Delayed Teriparatide | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.0 (8.660) | 69.8 (8.085) | 74.2 (9.094)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Radiologic Evidence of Bone Healing
Description: The radiologic indices of fracture healing included (1) cortical continuity on two of four cortices, (2) persistence of alignment, (3) decreased conspicuity of fracture line, and (4) increased callus formation. For each of these indices, healing was graded on a scale of 1 to 4 with 1 = no change (less than 25%), 2 = minimum healing (25-50%), 3 = moderate healing (50-75%), and 4 = complete healing (greater than 75%). A composite score was calculated by summing the subscale scores for the 4 indices. Composite score scale ranged from 4 to 16 with higher scores indicating more complete healing. The primary grading was performed by a radiologist with expertise in musculoskeletal radiology, then independently repeated by a second radiologist, both of whom were blinded to the study allocation.
Time Frame: 6, 12 months of treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Immediate Teriparatide | Delayed Teriparatide
Number analyzed (Participants) | 7 | 6
units on a scale
  6 mo | 12.6 (0.6) | 11.2 (1.3)
  12 mo | 15.4 (0.4) | 13.2 (1.2)

2. Primary Outcome: Radiologic Evidence of Healing
Description: Number of participants with persistence of alignment as determined by a radiologist.
Time Frame: at 10 weeks for immediate teriparatide group
Population: Based on orthopedic surgeons' assessment, x-rays were not deemed necessary in over 30% of patients at week 10. Results presented are for those who had x-rays at 10 weeks to assess persistence of alignment for safety purposes.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Teriparatide | Delayed Teriparatide
Number analyzed (Participants) | 5 | 4
Participants | 5 | 4

3. Secondary Outcome: Radiologic Healing
Time Frame: at 2, 6, 24, and 48 weeks
Population: Data not collected at 2 and 6 weeks. Twenty-Four week (6 months) data is presented in 6 month outcomes, and 48 week (12 months) data as 12 month outcomes (See primary outcomes section above).
Arm/Group | Immediate Teriparatide | Delayed Teriparatide
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Increased Bone Density
Description: Percent change in Bone Mineral Density (BMD) as assessed by dual x-ray absorptiometry (DXA) at the spine, contralateral hip, distal 1/3 radius, and femoral neck
Time Frame: at 6 and 12 months
Measure: Mean (Standard Error); unit: percentage change in BMD
Arm/Group | Immediate Teriparatide | Delayed Teriparatide
Number analyzed (Participants) | 7 | 6
percentage change in BMD
  Spine-PA (6 months) | 2.1 (1.5) | -0.6 (1.3)
  Spine-PA (12 months) | 2.8 (2.0) | 5.4 (2.8)
  Total Hip (6 months) | -1.6 (1.5) | -0.8 (0.7)
  Total Hip (12 months) | -0.3 (1.8) | 1.5 (2.7)
  Femoral Neck (6 months) | -1.8 (2.1) | -2.7 (1.0)
  Femoral Neck (12 months) | -2.5 (3.0) | -1.9 (3.6)
  Distal 1/3 Radius (6 months) | -0.6 (1.9) | -0.7 (1.1)
  Distal 1/3 Radius (12 months) | -1.9 (1.7) | -6.1 (2.1)

5. Secondary Outcome: Quality of Life Improvements
Description: Assessed by quality of life questionnaire (SF-36). There are 8 subscales each ranging from 0-100 with higher scores indicating better quality of life.
Time Frame: at 12 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Immediate Teriparatide | Delayed Teriparatide
Number analyzed (Participants) | 7 | 4
units on a scale
  Physical functioning | 49.3 (6.5) | 65.0 (20.3)
  Physical health limitations | 48.2 (9.1) | 68.8 (21.2)
  Emotional health limitations | 75.0 (9.1) | 72.9 (19.7)
  Energy/Fatigue | 54.5 (7.4) | 59.4 (15.0)
  Emotional well-being | 80.7 (4.1) | 70.0 (9.1)
  Social functioning | 92.9 (4.6) | 65.6 (23.6)
  Pain | 72.9 (9.7) | 59.4 (21.2)
  General health | 66.1 (6.2) | 67.2 (12.1)

6. Secondary Outcome: Difference in Biochemical Markers of Bone Turnover
Description: upfront therapy group compared to delayed therapy group and no therapy group
Time Frame: intervals over 12-18 months depending on treatment group
Population: Funding unavailable for sample analysis.
Arm/Group | Immediate Teriparatide | Delayed Teriparatide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Immediate Teriparatide | Delayed Teriparatide
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 3/7 | 2/6
Other Adverse Events (participants affected / at risk) | 5/7 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Teriparatide (N=7) | Delayed Teriparatide (N=6)
elective back surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Ewings Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Discovered prior to initiation of treatment with teritparatide
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) — Developed cellulitis at surgical site following repair of femur fracture
Abnormal coagulation profile (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hematoma (General disorders) | 1 (1) | 0 (0) — Hospitalized for incision and drainage of right hip hematoma at femoral surgical site
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Teriparatide (N=7) | Delayed Teriparatide (N=6)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
aphasia (Nervous system disorders) | 1 (1) | 0 (0)
myringotomy (Ear and labyrinth disorders) | 1 (1) | 0 (0)
arthralgias (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 1 (1) | 0 (0)
macular degeneration (Eye disorders) | 1 (1) | 0 (0)
cataract removal (Surgical and medical procedures) | 1 (2) | 0 (0)
deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
gingivitis (General disorders) | 0 (0) | 1 (1)
periodontal gum surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
allergic rhinitis (Immune system disorders) | 0 (0) | 1 (1)
coronary artery disease (Vascular disorders) | 0 (0) | 1 (1)
cardiac catheterization (Surgical and medical procedures) | 0 (0) | 1 (1)
dizziness (General disorders) | 0 (0) | 1 (1)
varicella zoster (Infections and infestations) | 0 (0) | 1 (1)
thigh pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No